CLINICAL TRIAL: NCT03962010
Title: A Phase 2, 12-Week, Double-Blind, Randomized, Parallel Group, Multi-Centre Study to Evaluate Efficacy and Safety of GX-G6 on Glycaemic Control Versus Placebo and Open-Label Dulaglutide in Patients With Uncontrolled Type 2 Diabetes Mellitus
Brief Title: A Phase 2, 12-Week, Double-Blind, Efficacy and Safety of GX-G6 in Patients With Uncontrolled Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GX-G6-002
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose level 1 (Experimental)
  Interventions: Drug: GX-G6
- Dose level 2 (Experimental)
  Interventions: Drug: GX-G6
- Dose level 3 (Experimental)
  Interventions: Drug: GX-G6
- Dose level 4 (Experimental)
  Interventions: Drug: GX-G6
- Placebo (Placebo Comparator)
  Interventions: Drug: Control
- Dulaglutide (Active Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: GX-G6 — long acting anti-diabetic drug
  Arms: Dose level 1; Dose level 2; Dose level 3; Dose level 4
Drug: Control — Control
  Arms: Dulaglutide; Placebo

SUMMARY:
GX-G6-002 is a Phase 2, 12-week, randomized, parallel group, multi-centre, double blind, placebo-controlled and an open-label active comparator study.

DETAILED DESCRIPTION:
This study aims to establish the dose-response relationship of 4 dose cohorts of GX-G6 compared with double-blind placebo. These treatment cohorts will also be compared with open-label active control.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of T2DM ≥ 6 months prior to screening
2. HbA1c level of 7-10% (inclusive)

Exclusion Criteria:

1. Have known type 1 diabetes mellitus (T1DM)
2. History of severe hypoglycaemia defined as ≥ 2 episodes of severe hypoglycaemia within 6 months prior to screening
3. Have had ≥ 2 episodes of ketoacidosis or hyperosmolar state/coma requiring hospitalization in the 6 months prior to screening
4. Has fasting serum TG ≥ 500 mg/dL or 9 mmol/L at screening.
5. Patients receiving lipid-lowering therapy must have been on the same dose of therapy for the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 12

IPD SHARING:
Plan to Share IPD: Undecided